CLINICAL TRIAL: NCT03764566
Title: Loneliness, Social Belonging, and Adverse Childhood Experiences: "Me and the Others: Expectations and Evaluation of Social Relationships"
Brief Title: Me and the Others: Expectations and Evaluation of Social Relationships
Status: Withdrawn | Type: Observational
Why Stopped: project has been cancelled
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GRK_B3
Record Dates: First submitted 2018-11-27; First posted 2018-12-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Life Change Events; Loneliness
Keywords: childhood adversities; childhood neglect; childhood abuse; rejection sensitivity; justice sensitivity; loneliness
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Trauma control group: Individuals with adverse childhood experiences (e.g.childhood abuse or neglect) will be included as the experimental group of participants. Individuals will fill out the designated questionnaires (e.g. Childhood Trauma Questionnaire, Rejection Sensitivity Questionnaire, Loneliness questionnaires), will participate in a multimodal emotion recognition experiment as well as a virtual reality (VR) task.
  Interventions: Behavioral: Questionnaires
- Healthy control group: Individuals with no trauma history will be added as the healthy control group of participants. Individuals will fill out the designated questionnaires (e.g. Childhood Trauma Questionnaire, Rejection Sensitivity Questionnaire, Loneliness questionnaires), will participate in a multimodal emotion recognition experiment as well as a virtual reality (VR) task.
  Interventions: Behavioral: Questionnaires
- Clinical control group: Individuals with Borderline Personality Disorder (BPD) will be added as a clinical control group. Individuals will fill out the designated questionnaires (e.g. Childhood Trauma Questionnaire, Rejection Sensitivity Questionnaire, Loneliness questionnaires), will participate in a multimodal emotion recognition experiment as well as a virtual reality (VR) task.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — The intervention will include the implication of related questionnaires, followed by a lab experiment for social belonging with multiple modalities. Participants will be shown pictures of different faces and asked to judge their feelings towards them. Further, a VR task will include finding the way through a virtual maze with the help of two virtual characters.
  Other Names: Multimodal emotion recognition task; Virtual maze task with the use of Virtual Reality (VR)

SUMMARY:
Chronic and pervasive loneliness has been identified as an important factor in the relationship between adverse childhood experiences (ACE) (e.g. abuse and neglect) and mental disorders. However, the mechanisms determining loneliness after ACE are still needed to be disentangled. Therefore, this study aims to investigate the differential effect of ACE on alterations in cognition and the link between ACE and loneliness with an emphasis on the effect of type and timing of ACE.

DETAILED DESCRIPTION:
With the rationale of the detrimental effects of loneliness on mental and physical health may be based on the interactions between genetic predispositions and social-environmental influences (e.g. ACE) via affecting neurobiological and cognitive processing, goals of this project are 1) characterization of loneliness to understand whether people suffer from mental/somatic disorders, feel lonelier and this effect is particularly strong in those with a history of ACE, 2) understanding the determinants of chronic loneliness by investigating certain personality dispositions such as rejection sensitivity and justice sensitivity, genetic predisposition for loneliness and social environments during childhood and adolescence and 3) inquiring into the social-cognitive correlates of these potential determinants in people's life today

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with and without adverse childhood experiences + clinical control group (i.e. individuals with borderline personality disorder)

Exclusion Criteria:

* A lifetime history of psychotic or bipolar I disorders, current pregnancy, history of organic brain disease, skull or brain damage, or severe neurological illnesses.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals who are German speaker, willing to participate in the study and meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-31 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
University of California, Los Angeles (UCLA) Loneliness Scale | 10 mins
  A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item on a scale from 1 (Never) to 4 (Often). Ratings are summed up by taking the reversed items into consideration.
Rejection Sensitivity Questionnaire (RSQ) | 10 mins
  Rejection Sensitivity Questionnaire will be used to measure the cognitive and affective components of the rejection experience, namely rejection expectancy and rejection concern. RSQ involves nine hypothetical interpersonal situations to measure how respondents would feel or think in stated situations. Items are answered on a 6-point Likert scale from 1= "very unconcerned" to 6= "very concerned" for the rejection concern and 1= "very unlikely" to 6= "very likely" for the rejection expectancy. By multiplying the results of the two levels, total rejection sensitivity score is calculated and higher scores indicate higher sensitivity to rejection.
Justice Sensitivity Inventory (JSI) | 10 mins
  JSI includes for questionnaire scales assessing victim, observer, beneficiary and perpetrator sensitivity on four subscales. Scores for each subscale range from 0 to 50 based on 10 items (6-point rating scale ranging from 0 to 5). Higher scores indicate a higher sensitivity to justice. JSI involves 4 each have 2 dimensions in terms of the applicability of the question for the self and the others.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Lis, PD Dr., Principal Investigator — Zentralinstitut für Seelische Gesundheit (ZI), Mannheim
Locations (1):
- Zentralinstitut für Seelische Gesundheit, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official website of the research training program that this study is a part of. — http://www.grk2350.de/